CLINICAL TRIAL: NCT00231595
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Response Study to Evaluate the Efficacy and Safety of Topiramate in the Prophylaxis of Migraine
Brief Title: A Study of the Efficacy and Safety of Topiramate in the Prevention of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003208
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Migraine; Common Migraine; Classic Migraine; Headache
Keywords: Migraine; Common Migraine; Classic Migraine; Headache; Topiramate; Prophylaxis; Prevention
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura; Migraine with Aura; Headache | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of three doses of topiramate (50 milligrams[mg], 100mg, and 200mg per day) compared with placebo in the prevention of migraine. The study will also assess the dose response relationship and the efficacy of treatment with topiramate versus placebo on Health-Related Quality of Life.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, multi-center study to evaluate the efficacy and safety of three different doses of topiramate (50mg, 100mg, and 200mg daily) in migraine prophylaxis. The study consists of five phases: Baseline (determination of whether patients meet the eligibility criteria and tapering of any migraine medication patients are already taking), Double-Blind (patients receive either 50 milligrams[mg], 100mg, 200mg of topiramate, or placebo), Blinded Transition Phase (doses of study medication are adjusted over 7 weeks in preparation for the Open-Label Extension Phase), Open-Label Extension Phase (patients continue the study medication in open-label manner for up to 6 months; doses are adjusted to maximize effectiveness and minimize side effects), Taper/Exit Phase (study medication is slowly discontinued over 2 weeks). The primary study hypothesis is that one or more of the three doses of topiramate (50, 100, 200 mg/day) will be superior to placebo in the prophylaxis of migraine based on the change in monthly (28 day) migraine period rate from the Prospective Baseline Period to the Double-Blind Phase. Topiramate tablets (50milligrams [mg], 100mg, 200mg, or placebo) taken by mouth as twice-daily regimen during the 26-week Double-Blind Phase. Doses are adjusted and continued during the 6 month Open-Label Extension Phase after which they are tapered over 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Medical history consistent with migraine with or without aura according to the International Headache Society (IHS) for at least 6 months prior to the study
* Between 3 to 12 migraine periods and no greater than 15 headache days (migraine and non-migraine) per month during the Baseline Phase
* No clinically significant abnormalities on neurological exams, electrocardiogram (ECG) or clinical laboratory test results at baseline
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Patients with headaches other than migraine
* Patients with episodic tension or sinus headaches
* Onset of migraine after age of 50 years
* Patients who have failed more than two adequate regimens for migraine prophylaxis
* Patients who overuse pain medications or certain other medications

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2001-03; Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Change in monthly (28 day) migraine period rate from the prospective baseline period to the double-blind phase.

SECONDARY OUTCOMES:
Proportion of patients responding to the treatment. Changes from baseline to the double-blind phase in number of monthly migraine attacks, monthly migraine days, number of days/month requiring rescue medication and Health-Related Quality of Life measures

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Brandes JL, Saper JR, Diamond M, Couch JR, Lewis DW, Schmitt J, Neto W, Schwabe S, Jacobs D; MIGR-002 Study Group. Topiramate for migraine prevention: a randomized controlled trial. JAMA. 2004 Feb 25;291(8):965-73. doi: 10.1001/jama.291.8.965. PMID 14982912